CLINICAL TRIAL: NCT07091058
Title: Health Outcomes Associated With Algal Blooms of Cyanobacteria and Red Tide in in Florida: Long-Term Health Impacts of Harmful Algal Bloom Exposure, Phase 2
Brief Title: Harmful Algal Blooms
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Collaborators: Florida Atlantic University (Other); Florida Department of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: STUDY00007298
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Red Tide
Keywords: algae; Cyanobacteria; red tide; cyanotoxin; Harmful Algal Blooms (HABs); microcystins; brevetoxin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Questionnaire A: Participants will be assigned to complete Questionnaire A based on if they are new or returning participants and on the status of bloom at consent.
- Questionnaire B: Participants will be assigned to complete Questionnaire B based on if they are new or returning participants and on the status of bloom at consent.

SUMMARY:
The purpose of this study is to compare the frequency of symptoms, exposure and health impacts in persons living in areas where they are exposed to bloom and non-bloom periods of cyanobacteria and red tide in Florida.

DETAILED DESCRIPTION:
Florida has experienced multiple harmful algal blooms during the past several years of two predominant types of Florida red tides occur in the Gulf of Mexico and are due to proliferation of the dinoflagellate Karenia brevis which produces a suite of highly irritative compounds known as brevetoxins. Human illness is primarily due to inhalation of aerosols, which results in a well-characterized syndrome of respiratory tract symptoms due to the irritative effects of brevetoxin.

The proposed study will utilize a case-control approach to compare symptom frequency during bloom and non-bloom period sampling to compare exposures and health impacts. In addition, for the exposed group, comparison of bloom cell density will be examined. As in our previous study, sampling locations will include Fort Myers region, Stuart, and communities around Lake Okeechobee (for example Clewiston and Indiantown). Continuing data collection sites will include: The Volunteers in Medicine Clinic (VIM) in Stuart, Public Health Department in Clewiston, Florida Public Works Department in Cape Coral, and FAU Clinical Research Unit in Boca Raton, FL.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* live, visit, and/ or work in the following Florida counties: Indian River, St. Lucie, Charlotte, Collier, Hendry, Hillsborough, Lee, Manatee, Martin, Monroe, Okeechobee, Palm Beach, Pasco, Pinellas, Indian River, and/or Sarasota
* able to read and understand English

Exclusion Criteria:

* unable to independently consent
* younger than 18 years old
* prisoner
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include up to 400 individuals who are 18yrs of age or older, visit, live or work in specific Florida counties and who read and understand English and consent to participation.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To correlate self- reported symptom occurrence with recreational/occupational cyanotoxin exposure (measured in air and water environmental samples) and cyanotoxin levels in blood, nasal swab | 2 years
  These data will be linked to determine if and how much contact the participant may have had with Florida waters, presence of cyanotoxin in the bio samples (blood, nasal swabs, and urine) and self-reported health issues to determine the impact of harmful algal blooms (HABs) on human health. In addition, this study will explore a potential link between self-reported COVID-19 exposure/infection and susceptibility to cyanotoxins and establish a HAB biorepository.

SECONDARY OUTCOMES:
Continue the study of previously enrolled cohort participants prospectively to determine whether long-term effects can be attributed to exposure to microcystins and brevetoxins (Florida Red Tide). | 1 year
  Previously enrolled cohort participants will be screened, consented and enrolled, complete a questionnaire, self- collect nasal swab and urine sample and collection of blood.
Recruit and establish new study participants on the West Coast of Florida (coastal Lee County) to further study the health effects of exposure to Red Tide. | 1 year
  New participants will be screened, consented and enrolled, complete a questionnaire, self- collect nasal swab and urine sample and collection of blood.
Apply novel approaches to measure biomarkers in samples included in the biobank repository and maintained in the FAU Health Clinical Research Unit using using logistic regression and Generalized Linear Mixed Models (GLMM). | 2 years
  Access is granted through our continued relationship with FAU and Dr. McFarland as Co-PI. The concentrations of inflammatory biomarkers will be compared between 30 participants reporting dry cough, and/or wheezy respirations and 30 who reported neither of these symptoms and for whom serum samples are stored in the biobank. The data will be analyzed using parametric statistics with adjustment for potential confounders. Statistical analyses of the relationships between environmental concentrations of HAB toxins and concentrations in human tissues will be performed initially using standard regression techniques. Multivariable modelling of the relationships between environmental concentrations, tissue concentrations, symptom frequency and biomarkers will be conducted using logistic regression and Generalized Linear Mixed Models (GLMM) as appropriate for the data form.
Analysis of data collected during our previous studies in 2016, 2018, and 2020-2023 to explore risk factors that potentially increase the susceptibility to the respiratory impacts of harmful algal bloom toxin exposure. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Koszalinski, PhD, MS, RN, FIEL, CRRN, FARN, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Multiple Locations, Florida, United States